CLINICAL TRIAL: NCT06624072
Title: Relative Bioavailability of Two Different Formulations of Nerandomilast and Investigation of the Food Effect on New Formulation Following Oral Administration in Healthy Adult Male and Female Subjects (an Open-label, Randomised, Single-dose, Three-way Crossover Trial)
Brief Title: A Study in Healthy People to Compare 2 Different Formulations of Nerandomilast Tablets When Taken With or Without Food
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1305-0029; 2024-511245-18-00 (Registry Identifier: CTIS registry); U1111-1304-2287 (Registry Identifier: WHO register - International Clinical Trials Registry Platform (ICTRP))
Record Dates: First submitted 2024-10-01; First posted 2024-10-02 (Actual); Results first posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Healthy
MeSH Terms: interventions — BI 1015550

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Nerandomilast (18 mg) in treatment sequence R-T1-T2 (Experimental): Participants first received a single oral dose of 1 tablet of 18 milligrams (mg) nerandomilast adult formulation in the fasted state (Reference treatment, R), followed by a single oral dose of 18 tablets of 1 mg nerandomilast pediatric formulation in the fasted state (Treatment, T1), and then 18 tablets of 1 mg of nerandomilast pediatric formulation in the fed state as a single oral dose (Treatment, T2).
  Treatments were separated by a wash-out period of at least 7 days and treatments were taken with 240 mL of water after an overnight fast of at least 10 hours (hrs) for R and T1, or after a high-fat, high-calorie breakfast for T2.
  Interventions: Drug: Nerandomilast 18 mg - adult formulation; Drug: Nerandomilast 1 mg - paediatric formulation
- Nerandomilast (18 mg) in treatment sequence T1-T2-R (Experimental): Participants first received a single oral dose of 18 tablets of 1 mg nerandomilast pediatric formulation in the fasted state (T1), followed by a single oral dose of 18 tablets of 1 mg nerandomilast pediatric formulation in the fed state (T2), and then a single oral dose of 18 mg of nerandomilast adult formulation in the fasted state (R).
  Treatments were separated by a wash-out period of at least 7 days and treatments were taken with 240 mL of water after an overnight fast of at least 10 hrs for R and T1, or after a high-fat, high-calorie breakfast for T2.
  Interventions: Drug: Nerandomilast 18 mg - adult formulation; Drug: Nerandomilast 1 mg - paediatric formulation
- Nerandomilast (18 mg) in treatment sequence T2-R-T1 (Experimental): Participants first received a single oral dose of 18 tablets of 1 mg nerandomilast pediatric formulation in the fed state (T2), followed by a single oral dose of 18 mg of nerandomilast adult formulation in the fasted state (R), and then a single oral dose of 18 tablets of 1 mg nerandomilast pediatric formulation in the fasted state (T1).
  Treatments were separated by a wash-out period of at least 7 days and treatments were taken with 240 mL of water after an overnight fast of at least 10 hrs for R and T1, or after a high-fat, high-calorie breakfast for T2.
  Interventions: Drug: Nerandomilast 18 mg - adult formulation; Drug: Nerandomilast 1 mg - paediatric formulation

INTERVENTIONS:
Drug: Nerandomilast 18 mg - adult formulation — BI 1015550, oral tablet
  Other Names: BI 1015550, JASCAYD®
Drug: Nerandomilast 1 mg - paediatric formulation — BI 1015550, oral tablet
  Other Names: BI 1015550, JASCAYD®

SUMMARY:
The main objective of this trial is to investigate two different formulations of nerandomilast and the effect of food on the pharmacokinetics of the new formulation following oral administration.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (blood pressure (BP), pulse rate (PR)), 12-lead electrocardiogram (ECG), and clinical laboratory tests
* Age of 18 to 55 years (inclusive)
* Body mass index (BMI) of 18.5 to 29.9 kg/m² (inclusive)
* Signed and dated written informed consent in accordance with ICH-GCP and local legislation prior to admission to the trial Further inclusion criteria apply.

Exclusion Criteria:

* Any finding in the medical examination (including BP, PR or ECG) deviating from normal and assessed as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 45 to 90 beats per minute (bpm)
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator Further exclusion criteria apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2024-10-15 (Actual); Primary Completion 2024-11-22 (Actual); Study Completion 2024-11-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Humanpharmakologisches Zentrum Biberach, Biberach, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial was an open-label, single dose, 3-way crossover design. Subjects were randomly allocated to one of 3 treatment sequences. Each subject participated in 3 treatment periods, receiving a single dose in each, with a washout period of at least 7 days between treatments.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Period: Treatment Period 1
Arm/Group | Nerandomilast (18 mg) in Treatment Sequence R-T1-T2 | Nerandomilast (18 mg) in Treatment Sequence T1-T2-R | Nerandomilast (18 mg) in Treatment Sequence T2-R-T1
Started | 5 | 5 | 5
Completed | 5 | 5 | 5
Not Completed | 0 | 0 | 0
Period: Washout Period 1 (7 days)
Arm/Group | Nerandomilast (18 mg) in Treatment Sequence R-T1-T2 | Nerandomilast (18 mg) in Treatment Sequence T1-T2-R | Nerandomilast (18 mg) in Treatment Sequence T2-R-T1
Started | 5 | 5 | 5
Completed | 5 | 5 | 4
Not Completed | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 1
Period: Treatment Period 2
Arm/Group | Nerandomilast (18 mg) in Treatment Sequence R-T1-T2 | Nerandomilast (18 mg) in Treatment Sequence T1-T2-R | Nerandomilast (18 mg) in Treatment Sequence T2-R-T1
Started | 5 | 5 | 4
Completed | 5 | 5 | 4
Not Completed | 0 | 0 | 0
Period: Washout Period 2 (7 days)
Arm/Group | Nerandomilast (18 mg) in Treatment Sequence R-T1-T2 | Nerandomilast (18 mg) in Treatment Sequence T1-T2-R | Nerandomilast (18 mg) in Treatment Sequence T2-R-T1
Started | 5 | 5 | 5
Completed | 5 | 5 | 5
Not Completed | 0 | 0 | 0
Period: Treatment Period 3
Arm/Group | Nerandomilast (18 mg) in Treatment Sequence R-T1-T2 | Nerandomilast (18 mg) in Treatment Sequence T1-T2-R | Nerandomilast (18 mg) in Treatment Sequence T2-R-T1
Started | 5 | 5 | 5
Completed | 5 | 5 | 5
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS): The treated set included all subjects who were treated with at least one dose of trial drug. The number of subjects reported in each arm represents the number of subjects who took the first treatment in the respective sequence.
Groups:
- Total: Total of all reporting groups
Arm/Group | Nerandomilast (18 mg) in Treatment Sequence R-T1-T2 | Nerandomilast (18 mg) in Treatment Sequence T1-T2-R | Nerandomilast (18 mg) in Treatment Sequence T2-R-T1 | Total
Number analyzed (Participants) | 5 | 5 | 5 | 15
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.2 (10.5) | 37.8 (10.1) | 39.8 (8.6) | 39.3 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 5 | 12
  Male | 1 | 2 | 0 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 5 | 5 | 15
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 5 | 5 | 5 | 15
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: AUC0-tz (Area Under the Concentration-time Curve of Nerandomilast in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point) for Treatment T1 vs Reference R
Description: AUC0-tz (area under the concentration-time curve of nerandomilast in plasma over the time interval from 0 to the last quantifiable data point) for Treatment T1 vs Reference R is reported. Geometric least square mean (adjusted geometric mean) and standard error (adjusted geometric standard error) were calculated using an analysis of variance (ANOVA) model on the logarithmic scale restricted to the data of interest for each comparison. The pharmacokinetic (PK) endpoints were log-transformed (natural logarithm) prior to fitting the ANOVA model. The model included the effect 'subjects within sequences' as random and the other effects of sequence, period and treatment were considered as fixed. These quantities were then back-transformed to the original scale to provide the point estimate and the 90% confidence interval (CI).
Time Frame: Within 3 hours (hrs) before and 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.5, 3, 4, 6, 8, 10, 12, 24, 34, 48, 58, 72, and 96 hrs after drug administration. For dosing after 58hrs, a tolerance of +/- 2 hrs was allowed.
Population: Pharmacokinetic (PK) parameter analysis set (PKS): This set included all subjects in the treated set (TS) who provided at least one PK endpoint that was defined as primary or secondary and was not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability. Thus, a subject was included in the PKS, even if he/she contributed only one PK parameter value for one period to the statistical assessment. Only participants with available data were analyzed.
Measure: Geometric Least Squares Mean (Standard Error); unit: hours*nanomoles/Liter (h·nmol/L)
Groups:
- Nerandomilast 18 mg Pediatric (Ped) Fasted State (Treatment T1): Participants received a single oral dose of 18 tablets of 1 mg nerandomilast pediatric formulation in the fasted state.
- Nerandomilast 18 mg Adult Fasted State (Reference R): Participants received a single oral dose of 1 tablet of 18 mg nerandomilast adult formulation in the fasted state.
Arm/Group | Nerandomilast 18 mg Pediatric (Ped) Fasted State (Treatment T1) | Nerandomilast 18 mg Adult Fasted State (Reference R)
Number analyzed (Participants) | 15 | 14
hours*nanomoles/Liter (h·nmol/L) | 2732.81 (NA) — Adjusted geometric standard error = 1.09 | 2647.2 (NA) — Adjusted geometric standard error = 1.09
Statistical Analysis 1: Comparison: Nerandomilast 18 mg Pediatric (Ped) Fasted State (Treatment T1) vs Nerandomilast 18 mg Adult Fasted State (Reference R); Ratio of adjusted geometric means was calculated using an analysis of variance (ANOVA) model on the logarithmic scale. The pharmacokinetic endpoints were log-transformed (natural logarithm) prior to fitting the ANOVA model. The model included the effect 'subjects within sequences' as random and the other effects of sequence, period and treatment were considered as fixed. These quantities were then back-transformed to the original scale; Test type: Other; Ratio of adjusted geometric means (T1/R) = 103.23, 90% CI 2-sided [97.31 to 109.52] — Ratio as percentage [%] Intra-individual geometric coefficient of variation (gCV) = 8.7%

2. Primary Outcome: AUC0-tz (Area Under the Concentration-time Curve of Nerandomilast in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point) for Treatment T2 vs T1
Description: AUC0-tz (area under the concentration-time curve of nerandomilast in plasma over the time interval from 0 to the last quantifiable data point) for Treatment T2 vs T1 is reported. Geometric least square mean (adjusted geometric mean) and standard error (adjusted geometric standard error) were calculated using an analysis of variance (ANOVA) model on the logarithmic scale restricted to the data of interest for each comparison. The pharmacokinetic (PK) endpoints were log-transformed (natural logarithm) prior to fitting the ANOVA model. The model included the effect 'subjects within sequences' as random and the other effects of sequence, period and treatment were considered as fixed. These quantities were then back-transformed to the original scale to provide the point estimate and the 90% CI.
Time Frame: as for outcome 1
Population: Pharmacokinetic (PK) parameter analysis set (PKS): This set included all subjects in the treated set (TS) who provided at least one PK endpoint that was defined as primary or secondary and was not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability. Thus, a subject was included in the PKS, even if he/she contributed only one PK parameter value for one period to the statistical assessment.
Measure: Geometric Least Squares Mean (Standard Error); unit: hours*nanomoles/Liter (h·nmol/L)
Groups:
- Nerandomilast 18 mg Ped Fed State (Treatment T2): Participants received a single oral dose of 18 tablets of 1 mg nerandomilast pediatric formulation in the fed state.
- Nerandomilast 18 mg Ped Fasted State (Treatment T1): Participants received a single oral dose of 18 tablets of 1 mg nerandomilast pediatric formulation in the fasted state.
Arm/Group | Nerandomilast 18 mg Ped Fed State (Treatment T2) | Nerandomilast 18 mg Ped Fasted State (Treatment T1)
Number analyzed (Participants) | 15 | 15
hours*nanomoles/Liter (h·nmol/L) | 2611.55 (NA) — Adjusted geometric standard error = 1.09 | 2732.81 (NA) — Adjusted geometric standard error = 1.09
Statistical Analysis 1: Comparison: Nerandomilast 18 mg Ped Fed State (Treatment T2) vs Nerandomilast 18 mg Ped Fasted State (Treatment T1); [analysis description as in outcome 1, analysis 1]; Test type: Other; Ratio of adjusted geometric means, T2/T1 = 95.56, 90% CI 2-sided [89.37 to 102.18] — Ratio as percentage [%] Intra-individual geometric coefficient of variation (gCV) = 10.3%

3. Primary Outcome: Cmax (Maximum Measured Concentration of Nerandomilast in Plasma) for Treatment T1 vs Reference R
Description: Cmax (maximum measured concentration of nerandomilast in plasma) for Treatment T1 vs Reference R is reported. Geometric least square mean (adjusted geometric mean) and standard error (adjusted geometric standard error) were calculated using an analysis of variance (ANOVA) model on the logarithmic scale restricted to the data of interest for each comparison. The pharmacokinetic (PK) endpoints were log-transformed (natural logarithm) prior to fitting the ANOVA model. The model included the effect 'subjects within sequences' as random and the other effects of sequence, period and treatment were considered as fixed. These quantities were then back-transformed to the original scale to provide the point estimate and the 90% CI.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Least Squares Mean (Standard Error); unit: nanomoles/Liter (nmol/L)
Arm/Group | Nerandomilast 18 mg Ped Fasted State (Treatment T1) | Nerandomilast 18 mg Adult Fasted State (Reference R)
Number analyzed (Participants) | 15 | 14
nanomoles/Liter (nmol/L) | 501.74 (NA) — Adjusted geometric standard error = 1.10 | 480.85 (NA) — Adjusted geometric standard error = 1.10
Statistical Analysis 1: Comparison: Nerandomilast 18 mg Ped Fasted State (Treatment T1) vs Nerandomilast 18 mg Adult Fasted State (Reference R); [analysis description as in outcome 1, analysis 1]; Test type: Other; Ratio of adjusted geometric means, T1/R = 104.34, 90% CI 2-sided [91.00 to 119.65] — Ratio as percentage [%] Intra-individual geometric coefficient of variation (gCV) = 20.4%

4. Primary Outcome: Cmax (Maximum Measured Concentration of Nerandomilast in Plasma) for Treatment T2 vs T1
Description: Cmax (maximum measured concentration of nerandomilast in plasma) for Treatment T2 vs T1 is reported. Geometric least square mean (adjusted geometric mean) and standard error (adjusted geometric standard error) were calculated using an analysis of variance (ANOVA) model on the logarithmic scale restricted to the data of interest for each comparison. The pharmacokinetic (PK) endpoints were log-transformed (natural logarithm) prior to fitting the ANOVA model. The model included the effect 'subjects within sequences' as random and the other effects of sequence, period and treatment were considered as fixed. These quantities were then back-transformed to the original scale to provide the point estimate and the 90% CI.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Least Squares Mean (Standard Error); unit: nanomoles/Liter (nmol/L)
Arm/Group | Nerandomilast 18 mg Ped Fed State (Treatment T2) | Nerandomilast 18 mg Ped Fasted State (Treatment T1)
Number analyzed (Participants) | 15 | 15
nanomoles/Liter (nmol/L) | 344.76 (NA) — Adjusted geometric standard error = 1.07 | 501.74 (NA) — Adjusted geometric standard error = 1.07
Statistical Analysis 1: Comparison: Nerandomilast 18 mg Ped Fed State (Treatment T2) vs Nerandomilast 18 mg Ped Fasted State (Treatment T1); [analysis description as in outcome 1, analysis 1]; Test type: Other; Ratio of adjusted geometric means, T2/T1 = 68.71, 90% CI 2-sided [61.23 to 77.11] — Ratio as percentage [%] Intra-individual geometric coefficient of variation (gCV) = 17.9%

5. Secondary Outcome: AUC0-∞ (Area Under the Concentration-time Curve of Nerandomilast in Plasma Over the Time Interval From 0 Extrapolated to Infinity) for Treatment T1 vs Reference R
Description: AUC0-∞ (area under the concentration-time curve of nerandomilast in plasma over the time interval from 0 extrapolated to infinity) for Treatment T1 vs Reference R is reported. Geometric least square mean (adjusted geometric mean) and standard error (adjusted geometric standard error) were calculated using an analysis of variance (ANOVA) model on the logarithmic scale restricted to the data of interest for each comparison. The pharmacokinetic (PK) endpoints were log-transformed (natural logarithm) prior to fitting the ANOVA model. The model included the effect 'subjects within sequences' as random and the other effects of sequence, period and treatment were considered as fixed. These quantities were then back-transformed to the original scale to provide the point estimate and the 90% CI.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Least Squares Mean (Standard Error); unit: hours*nanomoles/Liter (h·nmol/L)
Arm/Group | Nerandomilast 18 mg Pediatric (Ped) Fasted State (Treatment T1) | Nerandomilast 18 mg Adult Fasted State (Reference R)
Number analyzed (Participants) | 15 | 14
hours*nanomoles/Liter (h·nmol/L) | 2748.78 (NA) — Adjusted geometric standard error = 1.09 | 2667.20 (NA) — Adjusted geometric standard error = 1.09
Statistical Analysis 1: Comparison: Nerandomilast 18 mg Pediatric (Ped) Fasted State (Treatment T1) vs Nerandomilast 18 mg Adult Fasted State (Reference R); [analysis description as in outcome 1, analysis 1]; Test type: Other; Ratio of adjusted geometric means, T1/R = 103.06, 90% CI 2-sided [97.22 to 109.25] — Ratio as percentage [%] Intra-individual geometric coefficient of variation (gCV) = 8.6%

6. Secondary Outcome: AUC0-∞ (Area Under the Concentration-time Curve of Nerandomilast in Plasma Over the Time Interval From 0 Extrapolated to Infinity) for Treatment T2 vs T1
Description: AUC0-∞ (area under the concentration-time curve of nerandomilast in plasma over the time interval from 0 extrapolated to infinity) for Treatment T2 vs T1 is reported. Geometric least square mean (adjusted geometric mean) and standard error (adjusted geometric standard error) were calculated using an analysis of variance (ANOVA) model on the logarithmic scale restricted to the data of interest for each comparison. The pharmacokinetic (PK) endpoints were log-transformed (natural logarithm) prior to fitting the ANOVA model. The model included the effect 'subjects within sequences' as random and the other effects of sequence, period and treatment were considered as fixed. These quantities were then back-transformed to the original scale to provide the point estimate and the 90% CI.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Least Squares Mean (Standard Error); unit: hours*nanomoles/Liter (h·nmol/L)
Arm/Group | Nerandomilast 18 mg Ped Fed State (Treatment T2) | Nerandomilast 18 mg Ped Fasted State (Treatment T1)
Number analyzed (Participants) | 15 | 15
hours*nanomoles/Liter (h·nmol/L) | 2631.39 (NA) — Adjusted geometric standard error = 1.09 | 2748.78 (NA) — Adjusted geometric standard error = 1.09
Statistical Analysis 1: Comparison: Nerandomilast 18 mg Ped Fed State (Treatment T2) vs Nerandomilast 18 mg Ped Fasted State (Treatment T1); [analysis description as in outcome 1, analysis 1]; Test type: Other; Ratio of adjusted geometric means, T2/T1 = 95.73, 90% CI 2-sided [89.47 to 102.42] — Ratio as percentage [%] Intra-individual geometric coefficient of variation (gCV) = 10.4%

ADVERSE EVENTS:
Time Frame: Adverse events: From intake of trial medication till end of the residual effect period (REP), up to 7 days for each treatment. All-Cause Mortality: Up to 7 days (REP) for each treatment (R, T1, T2), then follow-up (13 days), up to a total of 34 days.
Description: Treated set (TS): The treated set included all subjects who were treated with at least one dose of trial drug. The treated set was used for safety analyses.
Arm/Group | Nerandomilast 18 mg Adult Fasted State (Reference R) | Nerandomilast 18 mg Ped Fasted State (Treatment T1) | Nerandomilast 18 mg Ped Fed State (Treatment T2)
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 6/14 | 11/15 | 7/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nerandomilast 18 mg Adult Fasted State (Reference R) (N=14) | Nerandomilast 18 mg Ped Fasted State (Treatment T1) (N=15) | Nerandomilast 18 mg Ped Fed State (Treatment T2) (N=15)
Abdominal distension (Gastrointestinal disorders) | 0 | 2 | 1
Constipation (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 2 | 2
Vomiting (Gastrointestinal disorders) | 0 | 0 | 2
Fatigue (General disorders) | 1 | 0 | 0
Peripheral swelling (General disorders) | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Dizziness (Nervous system disorders) | 2 | 0 | 0
Headache (Nervous system disorders) | 4 | 7 | 6
Paraesthesia (Nervous system disorders) | 0 | 1 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 1 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Haematoma (Vascular disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2025-04-11): https://cdn.clinicaltrials.gov/large-docs/72/NCT06624072/Prot_000.pdf
  • Statistical Analysis Plan (2025-01-17): https://cdn.clinicaltrials.gov/large-docs/72/NCT06624072/SAP_001.pdf